CLINICAL TRIAL: NCT04744701
Title: A Comparison of Laboratory APTT Testing Versus Point of Care (Bedside) Activated Partial Thromboplastin Time (APTT) Testing in the Paediatric Intensive Care Population: An Assessment of Accuracy, Time Efficiency, and Cost-effectiveness
Brief Title: A Comparison of Laboratory Versus Point of Care (Bedside) APTT Testing
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Dr Tim Lee, Consultant in Paediatric Respiratory Medicine, University of Leeds
Other Study IDs: 239600
Record Dates: First submitted 2021-01-28; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Critical Care; Child
Keywords: Thromboplastin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Hemochron Signature Elite Whole Blood Microcoagulation System — Bedside test of Activated Partial Thromboplastin Time

SUMMARY:
The overall aim of the study is to determine whether point-of-care (bedside) Activated Partial Thromboplastin Time (APTT) testing would be better than laboratory APTT testing in the PICU population (restricted to children under 16 years of age).

DETAILED DESCRIPTION:
The overall aim of the study is to determine whether point-of-care (bedside) Activated Partial Thromboplastin Time (APTT) testing would be better than laboratory APTT testing in the PICU population (restricted to children under 16 years of age). To do this the investigators need to compare both forms of testing in the following areas:

1. Accuracy - using laboratory results as our control the investigators want to ascertain how reliable Point-of-care (bedside) testing with the Hemochron Signature Elite is by comparing paired samples. The Hemochron Signature Elite Whole Blood Microcoagulation System is a battery-operated, hand-held instrument that performs individual point-of-care coagulation tests, including APTT, on fresh or citrated whole blood. The Hemochron Signature Elite instrument is CE marked and complies with multiple safety standard requirements and directives. The investigators know that the Hemochron Signature Elite is not 100% accurate compared to the laboratory but the degree of inaccuracy, particularly in the paediatric population is not clear, if within acceptable & predictable limits the investigators would still be able to use this in clinical practice.
2. Time efficiency - in view of the fact the Hemochron Signature Elite is on PICU, results from this will be almost immediately available. The investigators then want to measure exactly how long it takes from the moment the laboratory sample is taken for the results to be available.
3. Cost-effectiveness - the investigators want to compare the costs of these two types of testing in detail, including costs for the Hemochron Signature Elite machine, Hemochron Signature Elite cuvettes, laboratory Clotting Screen bottles, laboratory Clotting Screen analysis, and maintaining the two different types of equipment. The investigators will also take into account any other regular costs (e.g. porters to take samples to the laboratory when the pod system is down). The investigators plan on seeking assistance from senior paediatric colleagues with more experience of health economics in doing a costs minimisation analysis

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Paediatric Intensive Care Unit under the age of 16 years

Exclusion Criteria:

-

Max Age: 15 Years | Sex: All
Age Groups: Child
Study Population: Patients admitted to Paediatric Intensive Care Unit under the age of 16 years
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of APTT result (measured in seconds) provided by Hemochron Signature Elite compared to standard laboratory APTT value as gold standard (measured in seconds) on paired samples, using Pearson Correlation | 6 hours
  APTT measured on fresh whole blood using Hemochron Signature Elite, the device converts this to a plasma equivalent value for clinical use, reported in seconds. The gold standard laboratory assay in our Trust uses ACL Top 750 Analyser, with APTT reported in seconds. Pearson Correlation Co-efficient will be used to determine level of agreement.

SECONDARY OUTCOMES:
Mean time efficiency of Hemochron Signature Elite to provide APTT result (measured in minutes till APTT result being available), compared to the mean time taken (in minutes) for the standard laboratory measure of APTT result to become available. | 6 hours
  Investigators will calculate the mean time difference between results being obtained using Hemochron Signature Elite point of care (bedside) testing using the time recorded on the data collection sheet and comparing this with the mean time the results were released by the standard hospital laboratory which is stated on the hospital results server. The laboratory staff will be blinded to ensure the timings are a genuine reflection of standard care within the hospital. Time taken for each method of APTT measurement will be measured from the moment the samples are obtained from participants until the result becomes available. Mean time taken by each method across all participants will be compared.
Cost effectiveness (in £ GBP) of Hemochron Signature Elite point of care APTT testing compared to standard laboratory measurement of APTT. This will be reported as overall mean cost (in £ GBP) to provide 1 APTT result using each system, for comparison. | 1 day
  Costs will be determined by combining the fixed costs such as the costs of analyzers, quality control testing, cuvettes and sampling equipment with the variable costs such as utilisation of porters to transport samples when the air-tube system is not working. Costs related to the Hemochron Signature Elite will be as per the manufacturer's price list. The cost of routine laboratory testing will be obtained from the Hospital pathology services management team

CONTACTS AND LOCATIONS:
Overall Officials: Tim Lee, MD, PhD, Principal Investigator — University of Leeds
Locations (1):
- Leeds Children's Hospital, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No